CLINICAL TRIAL: NCT00903279
Title: Treatment of Patients Colonized With Methicillin-Resistant Staphylococcus Aureus Prior to Bone and Joint Surgery (TOPS-MRSA)
Brief Title: Treatment of Patients Colonized With Methicillin-Resistant Staphylococcus Aureus Prior to Bone and Joint Surgery
Acronym: TOPS-MRSA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Bay Pines VA Healthcare System (U.S. Federal Agency)
Responsible Party: David P. Johnson, MD, Bay Pines VAHCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOPS2009
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2009-05

CONDITIONS: Orthopedic Procedures; Methicillin-resistant Staphylococcus Aureus
Keywords: MRSA colonization; Orthopedic Surgery; Altabax; Placebo
MeSH Terms: interventions — retapamulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Altabax (Experimental)
  Interventions: Drug: Altabax (retapamulin)

INTERVENTIONS:
Drug: Placebo — Placebo will be administered intranasally an amount approximating 0.25 ml will be applied to each nasal vestibule by sterile cotton applicator in the evening prior to surgery and immediately on call on the day of surgery.
  Arms: Placebo
Drug: Altabax (retapamulin) — Retapamulin 1% ointment will be administered intranasally an amount approximating 0.25 ml will be applied to each nasal vestibule by sterile cotton applicator in the evening prior to surgery and immediately on call on the day of surgery.
  Other Names: Retapamulin
  Arms: Altabax

SUMMARY:
The investigators anticipate that utilization of retapamulin preoperatively will eliminate MRSA colonization among patients who are colonized in their nares.

DETAILED DESCRIPTION:
Enhanced characterization of MRSA strains carried by patients and their eradication prior to surgery will significantly reduce healthcare costs to the VA by reducing the number of MRSA positive patients who need to be isolated and or closely monitored, and allow healthcare providers to better predict the patient's requirements. In addition, the application of molecular methods will facilitate faster tracking of MRSA postoperative infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted for an orthopedic surgical procedure
* All patients will be screened and admitted to the study prior to surgery regardless of eventual culture results for MRSA

Exclusion Criteria:

* Pregnancy
* Serious systemic illness due to renal, cardiac or hepatic disease
* Inability to complete follow-up assessments
* Allergy or intolerance to retapamulin
* BMI > 30
* Uncontrolled diabetes, severe anemia, thrombocytopenia or an underlying hematopoietic disorder or malignancy
* Patients with serious life-threatening illnesses and those with terminal illness not expected to survive for two years or more will not be enrolled
* Antibiotics administered during the course of the study will be recorded (name, dose and dates)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy of Retapamulin 1% ointment in eliminating patients MRSA colonization | 30 days

SECONDARY OUTCOMES:
Identify a predominant clone among the MRSA isolates in this study | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzane Silbert, PhD, Study Director — Bay Pines VAHCS
Locations (1):
- Bay Pines VAHCS, Bay Pines, Florida, United States